CLINICAL TRIAL: NCT06160856
Title: Correlation of Ultrasonography Indices of Venous Congestion With Intra-abdominal Pressure in ICU Patients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Kyriakos K. Trigkidis, Dr, National and Kapodistrian University of Athens
Other Study IDs: 35656
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Intra-Abdominal Hypertension; Venous Congestion
MeSH Terms: conditions — Intra-Abdominal Hypertension; Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal intra-abdominal pressure
  Interventions: Diagnostic Test: Abdominal ultrasound
- Elevated intra-abdominal pressure
  Interventions: Diagnostic Test: Abdominal ultrasound

INTERVENTIONS:
Diagnostic Test: Abdominal ultrasound — Measurement of venous congestion in abdominal target-organs (liver, kidneys) by calculating VExUS score
  Other Names: VExUS score calculation

SUMMARY:
The goal of this prospective observational study is to examine the potential association between intra-abdominal pressure and venous congestion as assessed by abdominal ultrasound, in critically ill patients in the Intensive Care Unit (ICU).

The main question it aims to answer is whether there is association between intra-abdominal pressure and Venous Excess Ultrasound (VExUS) score.

Participants will be sonographically assessed and their intra-abdominal pressure measured once within the first 3 days of ICU admission.

ELIGIBILITY:
Inclusion Criteria:

* Intubated ICU patients on controlled mechanical ventilation, receiving sedation. Patients must have urethral catheter in place.

Exclusion Criteria:

* age < 18 year old
* pregnancy / lactation
* primary liver disease (hepatic cirrhosis, hepatic space-occupying lesions, Budd-Chiari syndrome, portal vein thrombosis) or hepatic surgery
* end stage renal failure or on chronic dialysis
* non-intubated patients or intubated patients on non-controlled mechanical ventilation mode
* absence of urethral catheter, presence of suprapubic catheter, continuous bladder irrigation
* poor abdominal echogenicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients admitted in a 31-bed University-affiliated general ICU in a tertiary hospital (Evangelismos General Hospital, Athens, Greece). The ICU admitts both medical and surgical patients.
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
VExUS score difference between the 2 study groups (normal and elevated intra-abdominal pressure) | 01.12.2023 - 01.08.2024

IPD SHARING:
Plan to Share IPD: Undecided